CLINICAL TRIAL: NCT04899323
Title: Compares Changes in Pulmonary ITV Secondary to Vascular Filling to Reference Values Represented by Changes in Subaortic ITV in the Management of Sepsis in the Emergency Department.
Brief Title: Correlation of Aortic Versus Pulmonary ITV in Response to Vascular Filling
Acronym: CIAOP
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC21_0026
Record Dates: First submitted 2021-05-19; First posted 2021-05-24 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Sepsis With Hemodynamic Instability
Keywords: Aortic ITV; Pulmonary ITV; Cardiac ultrasound; Hemodynamic ultrasound; Vascular filling; Sepsis; Emergency medicine; Recommendations
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: Perform a 250cc vascular filling over 10 minutes and then perform a cardiac ultrasound. Repeat the vascular filling followed by the ultrasound as long as the patient is responsive.

SUMMARY:
This is a multicenter study conducted in the emergency department of the Nantes University Hospital and the Confluent Private Hospital, over a period of 5 months, based on hemodynamic ultrasound.

For each patient admitted to an emergency department with a sepsis syndrome requiring vascular filling, the pulmonary ITV and the aortic ITV were measured at each phase of vascular filling.

This is a non-interventional study, the management of patients will not differ from usual practices and vascular filling should not be delayed in any case. Emergency doctors who are already experts in ultrasound, monitoring vascular filling by measuring the aortic ITV, will have to measure the pulmonary ITV after each filling of 250cc of Ringer's Lactate in 10 minutes with a limited amount of time.

The evolution of ITV measurements and vital parameters should be recorded for each patient.

In order to ensure quality, the emergency doctors will first receive a short training (presentation of the study and review of the measurements requested). In addition, measurement records will be analyzed at random.

At the end of this study, the correlation between the variation of the aortic and pulmonary ITV could be compared. The objective would be to promote the monitoring of these unstable patients via the pulmonary ITV. This measurement would be easier to perform than the aortic ITV, which is currently only performed by emergency doctors who are experts in hemodynamic ultrasound.

ELIGIBILITY:
Inclusion Criteria :

* Age> 18 years
* Patient with suspected infectious syndrome
* qSOFA >= 2
* Tachycardia>120 and/or PAS < 100mm Hg / MAP <60 mmHg

Exclusion Criteria :

* Atrial fibrillation arrhythmia
* Vascular filling > 500 ml before hemodynamic evaluation by echo cardiography
* Perfusion of catecholamine (norepinephrine, epinephrine, or dobutamine) at the time of inclusion in the study (before hemodynamic assessment by echo cardiography)
* Patient sedated and on positive pressure ventilation, including NIV
* Tamponade due to a compressive pericardial or pleural effusion
* Patient with known pre-capillary PAH > 50 mmHg PAPS
* Presence of suspected acute valvulopathy requiring immediate cardiological expertise
* Absence of an acoustic window allowing the evaluation of the aortic or pulmonary ITV
* Minor patients, adults under guardianship, protected persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major patients with sepsis requiring vascular filling
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Demonstration of a correlation between changes in pulmonary ITV secondary to vascular filling and reference values represented by changes in subaortic ITV. | 5 months
  Aortic ITV and pulmonary ITV

SECONDARY OUTCOMES:
Investigate whether pulmonary ITV is more feasible than aortic ITV. | 5 months
  Proportion of cases where Aortic ITV measurement is not feasible as opposed to pulmonary ITV.
Exploratory search for an indicator threshold for pulmonary ITV corresponding to the 10% threshold of aortic ITV (provided that pulmonary ITV and aortic ITV are correlated) | 5 months
  Pulmonary ITV and Aortic ITV

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, Loire-Atlantique, France